CLINICAL TRIAL: NCT06008431
Title: Modulating Brain Networks to Reduce Gait Variability in Older Adults at Risk of Falling
Brief Title: Non-invasive Brain Stimulation to Improve Unsteady Gait in Older Adults (StimGait)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hebrew SeniorLife (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Pro00057363; K01AG075252 (NIH)
Record Dates: First submitted 2023-08-18; First posted 2023-08-23 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-06

CONDITIONS: Fall; Gait, Unsteady; Mobility Limitation
Keywords: transcranial direct current stimulation (tDCS); transcranial electrical stimulation (tES); Non-invasive brain stimulation (NIBS); Falls; Gait Variability; Sustained Attention; Dorsal Attention Network; Default Network
MeSH Terms: conditions — Gait Disorders, Neurologic; Mobility Limitation | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- tDCS intervention (Experimental): Ten, once-daily, 20-min sessions of tDCS will be provided over two consecutive weeks.
  Interventions: Device: Transcranial direct current stimulation (tDCS) (active)
- Sham and then tDCS (Sham Comparator): Five, once-daily, 20-min sessions of sham in week one followed by five, once-daily, 20-min sessions of tDCS in week two.
  Interventions: Device: Transcranial direct current stimulation (tDCS) (active); Device: Transcranial direct current stimulation (tDCS) (Sham)

INTERVENTIONS:
Device: Transcranial direct current stimulation (tDCS) (active) — The tDCS montage is developed to modulate the functional connectivity between the dorsal attention network and the default network.
Device: Transcranial direct current stimulation (tDCS) (Sham) — The tDCS "Acti-" Sham montage is developed to recreate the cutaneous sensations associated with tDCS, yet essentially a null electrical field over the networks of interest.
  Arms: Sham and then tDCS

SUMMARY:
Walking is a complex and continuous task that entails repetitive motions of the body. Relatively high gait variability sensitively predicts falls and cognitive decline in older adults. Previous work has identified an unique brain network relationship linked to gait variability and its relevant cognitive function (i.e., sustained attention). This project aims to develop a non-invasive brain stimulation montage designed to modulate the shared brain networks dynamics and to demonstrate its effects on resting state functional connectivity, gait and cognitive performance in older adults at risk for falls.

DETAILED DESCRIPTION:
This is a randomized controlled trial to examine the efficacy of a non-invasive brain stimulation intervention of tDCS to improve unsteady gait in older adults. The investigators will enroll 30 older adults with elevated gait variability. Participants will be randomized into one of two arms: a) 10 sessions of tDCS and b) 5 sessions of sham stimulation followed by 5 sessions of tDCS. Participants will engage in a set of pre-intervention assessments, the brain stimulation intervention - consisting of 10, once-daily, 20-min stimulation sessions over a 2-week period, and a set of post-intervention assessments. This project is expected to demonstrate that tDCS can be used to reduce gait variability in older adults.

ELIGIBILITY:
Inclusion Criteria:

* Aged 65 and above.
* Ability to speak and read English.
* Ability to walk independently and continuously for at least 1 minute.
* Elevated gait variability as defined by a coefficient of variation (CoV) about average stride time larger and equal to 0.025 during straight-line walking at preferred speed.

Exclusion Criteria:

* More than mild cognitive impairment defined by a Montreal Cognitive Assessment (MoCA) score less than 18.
* Parkinson's disease, multiple sclerosis, stroke, active brain tumor, or other neurological disorders.
* Self-reported pain or lower extremity deformity that significantly disrupts walking.
* Contraindications to MRI or tDCS.
* An episode of acute illness or exacerbation of a diagnosis that requires hospitalization or active treatment within the past 3 months.
* Current treatment for congestive heart failure, angina, uncontrolled arrythmia, deep vein thrombosis, or other uncontrolled cardiovascular events.
* Myocardial infarction, coronary artery bypass grafting, angioplasty, or other cardiac conditions within the past 3 months,
* Active cancer for which chemo/radiation therapy is being received.
* Psychiatric co-morbidity including major depressive disorder, schizophrenia, psychosis, or other psychiatric illness.
* Recent use of any sedating medications (sedatives, anti-psychotics, hypnotics, anti-depressants) or change in medication within the previous month.
* Chronic vertigo or other diagnosed vestibular disorders.
* Legal blindness, visual impairments that cannot be corrected with glasses, contact lenses, medicine, or surgery.
* Those without WiFi access
* Those who do not plan to live in their current homes for the duration of the study

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 27 (Actual)
Dates: Start 2024-06-03 (Actual); Primary Completion 2025-11-20 (Actual); Study Completion 2025-11-20 (Actual)

PRIMARY OUTCOMES:
Gait variability | Baseline, Immediate post-intervention, 1 month follow up
  This measure is captured by both Mobility Lab (APDM Inc) and the smart phone App. Gait variability is defined as the coefficient of variation to validated stride times.

SECONDARY OUTCOMES:
Gait speed | Baseline, Immediate post-intervention, 1 month follow up
  This measure is captured by Mobility Lab (APDM InC). Gait speed id defined by the time one takes to walk a specified distance.
Dual-task gait performance | Baseline, Immediate post-intervention, 1 month follow up
  Participants will be asked to walk under two conditions: 1) walk at a comfortable, self-selected speed and 2) walk while counting backward by 1' or 3's from a random 3-digit number. Dual-task gait characteristics will be captured while the participants concurrently walk and count. We will further calculate the cost one takes to complete the dual-task walking from walking at a comfortable, self-selected speed.
Accuracy (d prime) on the gradual onset continuous performance task (gradCPT) | Baseline, Immediate post-intervention, 1 month follow up
  The gradCPT is a computer-based cognitive task designed to measure sustained attention. Accuracy (d prime) on the gradCPT can be derived from the gradCPT analysis tool box.

CONTACTS AND LOCATIONS:
Overall Officials: On-Yee Lo, Ph.D., Principal Investigator — Hinda and Arthur Marcus Institute for Aging Research, Hebrew SeniorLife
Locations (1):
- Hinda and Arthur Marcus Institute for Aging Research, Hebrew SeniorLife, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The prospective plan is to have data available in a data repository.
Supporting Information: Study Protocol, SAP
Time Frame: The data will be available when the data are unblinded.
Access Criteria: Depending on the repositories in which the data is held. Use of the data will be restricted by permission and appropriate human subjects review of the prospective project.